CLINICAL TRIAL: NCT05343234
Title: Drug Name Identification an Ignored Patient's Problem That Needs a Solution
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 0305534
Record Dates: First submitted 2022-04-17; First posted 2022-04-25 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Remember the Name of a Given Drug

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients receiving the placebo medication (Experimental): tree different placebo drugs with tree different names and symbols one will be given twice daily one once in the morning one once before bedtime
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — tree different placebo drugs with tree different names and scheduled will be given
  Other Names: placebo drugs

SUMMARY:
Each of the recruited patient was given 3 different placebo drugs with 3 different mad up names to be taken for one month with different regiments.

The drug name resembled a real drug but with enough difference to prevent the patient from trying to buy it as a safety precaution. The name was printed on the box in English and Arabic letters. The coloured shape was printed to 2x2 cm dimension.

After one month the participants were intervened by a doctor blinded to the study. The doctor asked about the drug history of the patient. If the participant could remember the drug name and its correct regiment the doctor documented that. if the patent failed to remember the correct name and its regiment then the doctor asked the patient to try and remember anything about the drug.

Then the patient would be asked about the symbol on the drug and was it helpful for him in any way.

DETAILED DESCRIPTION:
A scoring system was used to evaluate pateints memory of the drugs used 0- 3 0 is the minimal score and will be given if no recall of any drug name and 3 is the maximum score and will be given if the patient could remember the name of the tree drugs correctly.

The same scoring system was used for the symbols

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II patients

Exclusion Criteria:

* severe or life-threatening condition
* severe visual impairment
* mental or cognitive dysfunction

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2022-04-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
score for remembering the drug name | memory will be tested after one month from prescribing the drugs
  A scoring system was used to evaluate patients memory of the drugs name used 0- 3 0 is the minimal score and will be given if no recall of any drug name and 3 is the maximum score and will be given if the patient could remember the name of the tree drugs correctly.
score for remembering the drug symbol | memory will be tested after one month from prescribing the drugs
  A scoring system was used to evaluate patients memory of the drugs symbol used 0- 3 0 is the minimal score and will be given if no recall of any drug symbol and 3 is the maximum score and will be given if the patient could remember the symbol of the tree drugs correctly.

CONTACTS AND LOCATIONS:
Overall Officials: yasser M osman, Principal Investigator — Alexandria University
Locations (1):
- Alexandria university, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No